CLINICAL TRIAL: NCT01140308
Title: CoEnzyme Q10 in Statin Myopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1RC1AT005836-01 (NIH)
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Statin Myopathy
Keywords: Statin Myopathy; CoEnzyme Q10; CoQ10; Statin Myalgia
MeSH Terms: interventions — coenzyme Q10; Ubiquinone; Tuberculin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator): Simvastatin 20mg + Placebo
  Interventions: Drug: Placebo
- Co Q10 (Active Comparator): Simvastatin 20mg + CoQ10
  Interventions: Drug: CoEnzyme Q10

INTERVENTIONS:
Drug: CoEnzyme Q10 — Randomization to Treatment: Simvastatin 20mg + 600 mg CoQ10 (pill) Load Subjects for 2 weeks on Treatment (CoQ10) Eight weeks of Treatment
  Other Names: CoQ10; Ubiquinone; Q10; CoQ; Q; Ubidecarenone
  Arms: Co Q10
Drug: Placebo — Randomization to Treatment: Simvastatin 20mg + Placebo 600mg Load Subjects for 2 weeks on Treatment Eight weeks of treatment
  Other Names: Sugar pill
  Arms: Sugar Pill

SUMMARY:
Statins (such as simvastatin or Zocor) are the most effective and widely prescribed medications to lower cholesterol levels and reduce the frequency of heart attacks, cardiac deaths and strokes. Unfortunately, statins can cause muscle discomfort or pain called "myalgia" in patients treated with these drugs. These symptoms often cause patients who need these medications to stop taking the drug. The cause of statin muscle pain is not known, but it is thought that a reduction of a vitamin-like substance called Coenzyme Q10 (CoQ10) during statin treatment may play a role. CoQ10 is a vitamin like substance and is not a drug approved and regulated by the Food and Drug Administration (FDA). This study will look at the effects of CoQ10 supplements on individuals who develop muscle symptoms while on simvastatin.

The investigators hope to test the hypothesis that CoQ10 supplementation compared to placebo in patients with documented statin myalgia reduces the intensity of pain during statin treatment.

DETAILED DESCRIPTION:
Study Overview: We estimate, based on the calculations detailed below that 80 subjects with documented statin myalgia will be required to test our hypothesis. Consequently, 135 patients with statin myopathic complaints will be recruited from the Cholesterol Management Center at Hartford Hospital, newspaper and radio advertisements and contact with physicians' offices. Subjects will be withdrawn from all lipid lowering medications for at least 4 weeks. Subjects will then have serum measured for baseline lipids, liver, kidney, and thyroid function, creatine kinase (CK) and CoQ10 values and be randomized to treatment with simvastatin 20 mg daily or matching placebo for up to 2 months. Subjects will be called weekly to assess symptoms. Blood measurements will be repeated and treatment (simvastatin or placebo) will stopped after 2 months or after subjects have experienced muscle symptoms continuously for one week. After 4 weeks, subjects will cross over to the alternative placebo or simvastatin treatment and the monitoring and measurement process will be repeated. Those patients developing myalgia during statin treatment, but not during placebo, will enter the CoQ10 study, again after 4 weeks off treatment. These subjects will have serum lipids, liver, CK, vitamin D and CoQ10 levels measured, 4mL of blood sample will be stored for future white blood cell analysis and they will undergo tests of muscle performance and exercise capacity. They will then be randomized to placebo or CoQ10 treatment arms, "loaded" with placebo or CoQ10 to ensure adequate tissue levels for two weeks, and then retreated with simvastatin 20 mg daily. Subjects will be called weekly to inquire about muscle symptoms. Blood measurements will be repeated, another 4mL of blood sample will be stored for future white blood cell analysis and treatment (simvastatin/CoQ10 or simvastatin/placebo) will be stopped after 2 months or after subjects have experienced muscle symptoms continuously for one week. After 4 weeks subjects will cross over to the alternative simvastatin/CoQ10 or simvastatin/placebo treatment and the monitoring and measurement will be repeated. The primary endpoint will be the intensity of pain at eight weeks, or after subjects have had continuous symptoms for a week (or less in the case of intolerable symptoms), whichever comes first. We will also determine time in days to the onset of repeat myopathic symptoms and measure muscle performance including skeletal muscle strength and endurance and maximal aerobic exercise capacity using techniques used in our present NIH funded research project The Effect of Statins on Skeletal Muscle Function (R01 HL081893). We will measure muscle strength, endurance and aerobic capacity because weakness is a frequent, but largely unquantified, complaint among patients with statin myalgia and its prevention with CoQ10 is therefore important. Also, some investigators have reported changes in the rest and exercise respiratory exchange ratio (RER) with statin therapy implying an alteration in cellular substrate metabolism with statins that may be influenced by CoQ10 treatment.

Study Subjects: Subjects will be recruited from the Cholesterol Management Center, which sees approximately 20 new patients weekly, the majority of whom have statin myalgia and who are referred because of Dr. Thompson's expertise in this topic, via advertisements and by physician contact by mail and email informing them of the study. Subjects will be reimbursed $500 for their participation in the study.

Study Definition of Statin-Related Myopathic Complaints: Statin myopathic symptoms have been poorly defined in the medical literature. For the purpose of this study, subjects will be considered to have had prior statin related complaints and recruited for participation in the study if all of the following occur:

1. They developed new myalgia, cramps, or muscle aching during statin treatment;
2. The symptoms resolved within 4 weeks of stopping the statin. Subjects meeting these criteria will be recruited into the study. To ensure that only patients with documented statin myalgia are entered into the CoQ10 trial, all subjects with a history of statin myalgia will be treated for up to 8 weeks with simvastatin 20 mg daily or placebo in a double-blind, cross-over protocol.

Those developing statin myalgia only during simvastatin treatment will be advanced to the CoQ10 trial.

Throughout the study, subjects will be contacted by phone weekly to inquire about muscle complaints using the Brief Pain Inventory (Short Form) (BPI-SF) (18). Results will be recorded on paper forms and entered into the database. During the phone contacts, subjects with symptoms for statin myopathy will have a CK level determined within 72 hours and while on study drug. If the CK is > 10 times upper limits of normal (UNL), the standard diagnosis of myositis, and is unassociated with recent exercise, the drug will be stopped and the subject will undergo prompt repeat testing and be removed from the study. If the CK is < 10 UNL, the drug will be continued until the subject has had symptoms for 1 week to document that the symptoms are not transitory. After 1 week of persistent symptoms or as soon as possible if the patient has intolerable symptoms, the subject will undergo final testing and have completed the study. This reduces undue subject burden such that subjects do not have to maintain statin treatment for multiple weeks with pain symptoms. Subjects who do not report recurrent symptoms will be treated for 8 weeks, at which time they will undergo final testing and have completed the study.

Justification of Primary Endpoint: We will examine the ability of CoQ10 to reduce the intensity of pain because many patients would remain on statin therapy if the discomfort were tolerable. Consequently, increasing pain tolerability is a key clinical measure. We selected 8 weeks of therapy for the simvastatin vs placebo and CoQ10 vs placebo sections of the study because in the largest clinical study, the median time to onset of myalgia in statin naïve subjects was 1 month and statin rechallenge typically reproduces symptoms more rapidly. Consequently, most subjects with true statin myalgia will have clearly developed symptoms at or before 8 weeks, the point at which study procedures are completed, allowing us to accurately assess the impact of CoQ10 on muscle pain intensity. Except for chronic aspirin use, commonly recommended in patients at risk for heart disease, or in patients chronically using pain medications even off statin therapy, over the counter pain medication use for myalgic or myopathic symptoms will be prohibited during the study.

Study outline:

135 Subjects with Prior Statin Complaints:Stop Cholesterol Drugs for at least 4 Weeks

Run-In: Initial - Simvastatin or Placebo

1. Phlebotomy: Lipids1, ALT, creatinine, TSH, CK, CKMB, Vitamin D and CoQ10
2. Arterial Stiffness
3. FMD/Nitroglycerin administration
4. Simvastatin 20 mg for 8 weeks or Until Symptoms Persist for 1 Week or are Intolerable
5. Obtain lipids and CK

**4-week washout followed by crossover and repeat 1 - 5**

**4-Week Washout**

**100 Subjects Symptomatic on Statins Only(CoQ10 treatment phase)**:

1. Phlebotomy: Lipids, ALT, creatinine, CK, CKMB, Vitamin D and CoQ10, 4mL sample stored for future white blood cell analysis
2. Baseline Strength and Exercise Performance Testing, Accelerometer, Pain Questionnaire
3. Randomization to Treatment: Placebo or 600 mg CoQ10
4. Load Subjects for 2 weeks on Treatment

Simvastatin 20mg + Placebo (N=50) or Simvastatin 20mg + CoQ10 (N=50)

Weekly phone calls: Pain Questionaires

At 8 Weeks or Until Symptoms Persist 1 Week or are Intolerable:

1. Phlebotomy: Lipids, ALT, creatinine, CK, CKMB and CoQ10, Vitamin D, 4mL sample stored for future white blood cell analysis
2. Arterial stiffness
3. Strength and Exercise Performance Testing,Accelerometer, Pain Questionnaire

**4 week washout followed by crossover, repeat 1-4 and 1-3 above**

Weekly phone calls used to assess muscle symptoms and document myalgia

All visits include a Cognitive Failures Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* We will not exclude patients with diagnosed CAD, peripheral vascular disease or diabetes since these patients warrant aggressive lipid treatment, and would benefit from any intervention that increases their tolerance of statins. We do not consider it inappropriate or unethical to place such patients on placebo during the simvastatin vs placebo phase because these patients will have previously been documented to be intolerant of statins. All patients will be maintained on lipid lowering diets during the study.
* LDL Cholesterol Levels - LDL levels will not be a criterion for inclusion or exclusion from this study since all patients will have previously been deemed appropriate candidates for statin therapy by their physicians and because recent clinical trial results suggest that statins will be used in high risk individuals regardless of their pretreatment LDL-C values.
* Race - We will seek to recruit Caucasians, Hispanics and African American in accordance with their distributions in the study communities.
* CoQ10 Use - Subjects previously using supplemental CoQ10 must discontinue this supplementation for two months prior to entering the study.
* Diet - All subjects will be instructed in a standard lipid lowering diet and asked to maintain this throughout the 6 months of the study.

Exclusion Criteria:

* Subjects will be excluded if they have had cancer within 5 years of entry, have hepatic disease (ALT > 2 times normal) or renal disease (creatinine > 2 mg/L) since these patients may require more careful monitoring during the study and would be best managed in a totally clinical setting.
* Subjects presently treated with other medications known to alter statin metabolism (3)
* Subjects who cannot discontinue other lipid-lowering medications
* Subjects with hypo or hyper thyroidism defined as a TSH > 5 or <0.01 IU/L since these conditions are known to be associated with statin intolerance and muscle weakness, respectively
* Subjects with hepatic dysfunction evidenced by a baseline alanine aminotransferase (ALT) level > 2 UNL
* Subjects with renal dysfunction defined as a baseline creatinine > 2mg/dl;
* Subjects with physical disabilities prohibiting the strength and exercise performance measurements
* Subjects who regularly use corticosteroids or other drugs known to affects skeletal muscle metabolism or regularly have intramuscular injections that will affect CK levels.
* Women of child-bearing potential who do not use an effective birth-control technique.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
To test the hypothesis that CoQ10 supplementation compared to placebo in patients with documented statin myalgia reduces the intensity of pain during statin treatment. | We selected 8 weeks of therapy .
  Increasing pain tolerability is a key clinical measure. We selected 8 weeks of therapy for the simvastatin vs placebo and CoQ10 vs placebo sections of the study because in the largest clinical study, the median time toonset of mylagia in statin naïve subjects was 1 month (4) and statin rechallenge typically reproduces symptoms more rapidly(3). Consequently, most subjects with true statin myalgia will have clearly developed symptoms at or before 8 weeks, the point at which study procedures are completed, allowing us to accurately assess the impact of CoQ10 on muscle pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Thompson, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

REFERENCES:
- [Derived] Taylor BA, Lorson L, White CM, Thompson PD. Low vitamin D does not predict statin associated muscle symptoms but is associated with transient increases in muscle damage and pain. Atherosclerosis. 2017 Jan;256:100-104. doi: 10.1016/j.atherosclerosis.2016.11.011. Epub 2016 Nov 12. PMID 27993387
- [Derived] Taylor BA, Lorson L, White CM, Thompson PD. A randomized trial of coenzyme Q10 in patients with confirmed statin myopathy. Atherosclerosis. 2015 Feb;238(2):329-35. doi: 10.1016/j.atherosclerosis.2014.12.016. Epub 2014 Dec 17. PMID 25545331